CLINICAL TRIAL: NCT03976843
Title: A Phase II Multi-Institutional Trial to Evaluate Prostate Specific Membrane Antigen (PMSA)-Based PET Imaging of High Risk Prostate Cancer
Brief Title: Prostate Specific Membrane Antigen (PMSA)-Based PET Imaging of High Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Lantheus (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190104; 19-C-0104
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12-16

CONDITIONS: Prostate Cancer
Keywords: PSMA; PET agent; Prostatectomy; Progression Free Survival
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/18F-DCFPyL PET/CT + radical prostatectomy (Experimental): 18F-DCFPyL PET/CT with radical prostatectomy and lymphadenectomy
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-labeled agent that is a high affinity small molecule inhibitor of PSMA to detect prostate cancer via PET imaging

SUMMARY:
Background:

People with prostate cancer usually have their cancer imaged with a CT scan and bone scan. They then have their prostate gland removed. Researchers want to test a scan that might predict if prostate cancer will return after this surgery.

Objective:

To test if a PET/CT scan before the prostate gland is removed can predict if prostate cancer will return. Also, to test if this approach is better or worse than the usual approach for prostate cancer.

Eligibility:

Men ages 18 and older with prostate cancer that appears to be contained within the prostate but is at risk of having spread

Design:

Participants will be screened with:

* Medical history
* Blood tests
* CT and MRI scans: Participants will lie in a machine. The machine will take pictures of the body.
* Bone scan

Participants will have a radiotracer injected into a vein. They will have a PET/CT scan of their whole body 60-90 minutes later. During the scan, they will lie on their back and stay still.

Within 60 days after the scan, participants will have surgery. This will remove the prostate gland and lymph nodes around it. Some tissue will be used for genetic testing.

If the PET/CT scan suggests the cancer has spread, participants may need to have another biopsy within 60 days after the scan.

After surgery, participants will have follow-up visits for 5 years. They will have 5 visits the first year and 2 the second. Then they will have visits once a year.

If participants cancer returns, they will have repeat PET/CT scans.

DETAILED DESCRIPTION:
Background:

* About 30,000 men will die from prostate cancer in the US in 2018. The majority of these men originally presented with localized cancer.
* Treatment options for patients with high risk, localized disease typically involve radical prostatectomy (RP) or radiation therapy (RT) in combination with androgen deprivation therapy (ADT). Following RP, 70% of patients with high-risk disease will experience a biochemical recurrence at 5 years, and approximately 20% will die of their disease in 10-15 years, likely due to metastatic disease that was not detectable using conventional imaging (99mTc-methylene diphosphonate bone scan and X-ray computed tomography) at

the time of prostatectomy.

* Prostate-specific membrane antigen (PSMA) is commonly expressed in prostate cancers and is associated with biologic aggressiveness.
* The second generation, PET tracer 18F-DCFPyl binds to the enzymatic portion of PSMA. It exhibits high uptake in tumor and rapid washout in normal tissues leading to high tumor to background ratios and the possibility of detecting metastases when conventional imaging is negative.

Objective:

-To determine if patients with a preoperative 18F-DCFPyL PET/CT that is negative for metastases experience 5 year progression free survival (PFS) which is improved (40%) over that of historical data (30%) based on a general population of similar patients who have not undergone imaging with 18F-DCFPyL PET/CT

Eligibility:

* 18 years of age at the time of providing informed consent.

  * Patients must have histologically proven prostate adenocarcinoma confirmed by a CLIA certified laboratory
  * Eastern Cooperative Oncology Group (ECOG) performance status: <=2.
  * Must have prostate cancer with high risk features defined as:

    * Gleason 8 and higher OR
    * PSA > 20 ng/mL OR
    * Clinical stage T3a (i.e. likely extraprostatic extension on MRI) or T3b
  * Laboratory parameters:

    * Hemoglobin >= 9 g/dL
    * Leukocytes >=3,000/mcL
    * Platelets >=100,000/mcL
    * Total bilirubin <2 X normal institutional limits
    * AST(SGOT)/ALT(SGPT) <=3 X normal institutional limits
    * Creatinine <2 X normal institutional limits OR
    * eGFR >=50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (calculated via the MDRD equation)
  * Patients must be planning to undergo radical prostatectomy and lymphadenectomy regardless of findings on 18F-DCFPyL PET/CT.
  * Willingness and ability to undergo multiparametric prostate MRI and 18F-DCFPyL PET/CT

Design:

* This is an open-label, non-randomized, multi-center trial designed to evaluate the impact of 18F-DCFPyL PET/CT imaging on Progression-Free Survival at 5 years in patient with high risk localized prostate cancer.
* All subjects meeting eligibility criteria will undergo baseline assessments to include multiparametric MRI of the prostate, 99mTc-methylene diphosphonate bone scan and contrast-enhanced CT of the abdomen and pelvis.
* All subjects meeting eligibility criteria will undergo 18F-DCFPyL PET/CT.
* The study will enroll up to 200 patients from 7 centers. Up to 40 patients will be enrolled at NCI.
* All subjects will undergo radical prostatectomy and lymphadenectomy within 60 days following PET/CT imaging.
* Subjects will be evaluated at 6 weeks, at 3, 6, 9, 12, and 18 months, at 2, 3, 4, and 5 years post-prostatectomy to determine if there has been progression and to record details of subsequent treatment and response.
* 18F-DCFPyL PET/CT imaging will be repeated at the time of progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically proven prostate adenocarcinoma confirmed by a CLIA certified laboratory.
* Must have prostate cancer with high risk features defined as:

  * Gleason 8 and higher OR
  * PSA > 20 ng/mL OR
  * Clinical stage T3a (i.e. likely extraprostatic extension on MRI) or T3b
* Patients must be eligible for and must be planning to undergo radical prostatectomy and lymphadenectomy regardless of findings on 18F-DCFPyL PET/CT
* Men age greater than or equal to 18 years.
* ECOG performance status <2
* Patients must have adequate organ and marrow function as defined below:

  * Hemoglobin greater than or equal to 9 g/dL
  * leukocytes greater than or equal to 3,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin <2 X normal institutional limits
* AST(SGOT)/ALT(SGPT) less than or equal to 3 X normal institutional limits
* creatinine <2 X normal institutional limits

OR

eGFR greater than or equal to 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willingness and ability to undergo biopsy of radiotracer-avid lesion if feasible.
* Willingness and ability to undergo multiparametric prostate MRI and 18F-DCFPyL PET/CT

EXCLUSION CRITERIA:

* Any investigational agents in the past 28 days prior to enrollment.
* Clinical stage T4 (tumor invades adjacent structures except seminal vesicles).
* Distant metastatic disease on conventional imaging studies (computed tomography (CT)) of the abdomen and pelvis and bone scan. NaF PET/CT scan cannot substitute for a bone scan. Given lack of specificity of CT for lymph node metastases at lower thresholds, pelvic lymph nodes below 2 cm in the short axis are allowed.
* Any prior hormone therapy used to treat prostate cancer, except limited androgen receptor antagonist therapy, defined as less than or equal to 3 days of treatment. The medication must be discontinued within 5 half-lives of the compound prior to study entry.
* Any prior therapy for prostate cancer with surgery, radiation, and/or chemotherapy.
* Contraindication to MRI or PET:

  * Patients weighing more than weight limit for the scanner tables or unable to fit within the imaging gantry
  * Prior reaction to 18F-DCFPyL
  * Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic device that are not MRI compatible at 3 T
  * Severe claustrophobia unresponsive to oral anxiolytics
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other medical conditions deemed by the principal investigator (or associates) to make the subject unsafe/ineligible for the protocol procedures or for radical prostatectomy.
* A malignancy within the past 3 years for which prostatectomy is a contraindication.
* Radiotracer administered within 5 half-lives prior to the date of 18F-DCFPyL PET/CT imaging.
* PSMA-targeted imaging within 6 months with 18F-DCFPyL tracer prior to the date of 18F-DCFPyL PET/CT imaging. Participants can have PSMA targeted imaging with Gallium.
* Unable to refrain from fathering a child or donating sperm for 10 days after each 18FDCFPyL injection.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2027-11-19 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 weeks, 3,6,9,12, and 18 months, 2,3, and 4 years
  progression-free survival which is improved over that of historical data from a general population

SECONDARY OUTCOMES:
progression free survival | 6 weeks, 3,6,9,12, and 18 months, 2,3, and 4 years
  progression-free survival of patients with an 18F-DCFPyL PET/CT that is positive for metastases

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Brigham and Women s Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.@@@@@@Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI ETCTN Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0104.html
- See also: https://www.lantheus.com/ — https://www.lantheus.com/